CLINICAL TRIAL: NCT04268004
Title: Optimizing Fertility Preservation and Decision Quality in Male AYA With Cancer: A Family-centered Intervention
Brief Title: Fertility Preservation in Male AYA With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leena Nahata (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Leena Nahata, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00000849; K08CA237338 (NIH)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Infertility, Male
Keywords: Cancer; Fertility Preservation; Parenthood
MeSH Terms: conditions — Infertility, Male; Neoplasms

STUDY DESIGN:
Intervention Model Description: Families will be randomly assigned to receive standard care or to receive standard care plus the investigator's study intervention. All families will then be followed for a year to assess outcomes.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants, the interventionist, and research staff will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Control) (No Intervention): Participants will receive a standard of care fertility consult.
- FP Decision Tool and Discussion (Treatment) (Experimental): Participants will receive a standard of care fertility consult and will participate in a family-centered psychoeducational intervention consisting of completing a FP Decision Tool and participating in a guided discussion about responses and discrepancies identified in the FP Decision Tool.
  Interventions: Behavioral: FP Decision Tool and Discussion

INTERVENTIONS:
Behavioral: FP Decision Tool and Discussion — The intervention will be administered by a trained interventionist. The interventionist will administer the digital FP Decision Tool to families in the intervention arm. The tool asks questions examining each AYA's thoughts or feelings regarding parenthood and fertility preservation. The parent version asks the same questions, plus additional questions asking the parent to rate their son's feelings on certain topics (i.e., whether their son wants to have a child, whether their son would be as happy with an adopted child versus a biological child). Items are coded based on the domains of the Health Belief Model (perceived benefits, perceived barriers, perceived threats, self-efficacy, and cues to action). Items are scored and the trained interventionist will facilitate a guided discussion based on the family's responses and discrepancies.
  Arms: FP Decision Tool and Discussion (Treatment)

SUMMARY:
Very little is known about how medical providers can help adolescent and young adults (AYAs) and their caregivers make decisions about fertility preservation (sperm banking) before beginning cancer treatment. The purpose of this study is to see if having a guided conversation about fertility preservation increases preservation rates and/or satisfaction with the decision among AYA males with cancer. The primary hypothesis is that compared to standard of care control group (routine fertility consult at diagnosis, n=20), AYAs in the intervention arm (routine fertility consult at diagnosis + FP Decision Tool and Facilitated Conversation by trained interventionist) will have higher rates of FP uptake. The secondary hypothesis is that families in the intervention group will report better FP decision quality compared to those in the control arm.

DETAILED DESCRIPTION:
A rapidly growing population of male childhood cancer survivors are at risk for infertility and distress. As the number of male cancer survivors rises, it is essential to minimize treatment late effects. One of the most prevalent and significant complications among males is infertility, which can impair psychosocial development and reduce quality of life. National guidelines emphasize offering fertility preservation (FP) prior to initiation of cancer therapy, and sperm cryopreservation is an established and generally noninvasive FP method for pubertal males. Early research suggested only males receiving high doses of alkylating agents should bank sperm. However, variable sperm counts following equivalent doses of cyclophosphamide and scenarios in which patients have to move quickly from "low risk" treatments (which transiently impair sperm production) to "high risk" treatments, support the premise that all males receiving chemotherapy and/or gonadal radiation should consider FP at diagnosis. Despite studies showing ~50% of male childhood cancer survivors have fertility impairment, reports from many centers show only ~25% of pubertal males bank sperm prior to treatment. As survivors enter their reproductive years, many regret missed opportunities for FP and experience distress about potential infertility. Thus, interventions to improve FP uptake would have great potential for reproductive and psychological benefit.

Individual and family factors associated with sperm banking decisions remain poorly understood. Young age, cost, inadequate knowledge, and urgency to start treatment are common barriers to FP among AYA males with newly diagnosed cancer. As a result, most fertility counseling and FP interventions have targeted healthcare providers and systems or provider-patient interactions. While these are critical factors, less than half of male AYA advised about FP in a recent study actually banked sperm, indicating knowledge is not sufficient.

The purpose of this study is to test a decision tool and accompanying guided discussion as a method of improving decision making regarding FP, compared to a standard of care fertility consult.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 12-25 years
* Expected to have adjuvant therapy (chemotherapy and/or gonadal radiation) for newly diagnosed cancer
* Pubertal (at least Tanner stage 2-3, eligible for sperm banking as determined in the fertility consult)
* Proficient in English

Exclusion Criteria:

* Cognitive deficit that precludes completing measures
* Parents are non-English speaking

Ages: 12 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2025-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leena Nahata, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing individual participant data (IPD) with other researchers.

REFERENCES:
- [Background] Nahata L, Morgan TL, Lipak KG, Clark OE, Yeager ND, O'Brien SH, Whiteside S, Audino A, Quinn GP, Gerhardt CA. Perceptions of participating in family-centered fertility research among adolescent and young adult males newly diagnosed with cancer: A qualitative study. Pediatr Blood Cancer. 2019 Nov;66(11):e27966. doi: 10.1002/pbc.27966. Epub 2019 Aug 12. PMID 31407498
- [Background] Nahata L, Dattilo TM, Olsavsky AL, Lipak KG, Whiteside S, Yeager ND, Audino A, Klosky JL, Rausch J, Saraf A, O'Brien SH, Quinn GP, Gerhardt CA. Impact of a novel family-centered values clarification tool on adolescent sperm banking attempts at the time of a new cancer diagnosis. J Assist Reprod Genet. 2021 Jun;38(6):1561-1569. doi: 10.1007/s10815-021-02092-6. Epub 2021 Feb 10. PMID 33564937
- [Background] Theroux CI, Hill KN, Olsavsky AL, Klosky JL, Yeager ND, Audino A, O'Brien SH, Quinn GP, Gerhardt CA, Nahata L. Satisfaction with Fertility Preservation Decisions among Adolescent Males with Cancer: A Mixed Methods Study. Cancers (Basel). 2021 Jul 16;13(14):3559. doi: 10.3390/cancers13143559. PMID 34298773
- [Background] Nahata L, Olsavsky A, Dattilo TM, Lipak KG, Whiteside S, Yeager ND, Audino A, Rausch J, Klosky JL, O'Brien SH, Quinn GP, Gerhardt CA. Parent-Adolescent Concordance Regarding Fertility Perspectives and Sperm Banking Attempts in Adolescent Males With Cancer. J Pediatr Psychol. 2021 Oct 18;46(10):1149-1158. doi: 10.1093/jpepsy/jsab069. PMID 34333651
- [Background] Stanek C, Theroux CI, Olsavsky AL, Hill KN, Rausch JR, O'Brien SH, Quinn GP, Gerhardt CA, Nahata L. Study protocol for fertility preservation discussions and decisions: A family-centered psychoeducational intervention for male adolescents and emerging adults newly diagnosed with cancer and their families. PLoS One. 2022 Feb 16;17(2):e0263886. doi: 10.1371/journal.pone.0263886. eCollection 2022. PMID 35171948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited based on a medical chart review identifying patients with a new cancer diagnosis and/or through an automatic referral placed to the multidisciplinary Fertility and Reproductive Health Team following a new cancer diagnosis. Recruitment occurred at a single site (Nationwide Children's Hospital) in inpatient, outpatient, and remote settings. Recruitment occurred between February of 2021 and January of 2024.
Pre-assignment Details: No participants were excluded from the study after enrollment, but before assignment to groups.
Period: Overall Study
Arm/Group | Standard of Care (Control) | FP Decision Tool and Discussion (Treatment)
Started (Total number of participants (adolescents and caregivers) started) | 25 | 27
Adolescents Started | 10 | 9
Caregivers Started | 15 | 18
Adolescents Completed | 10 | 9
Caregivers Completed | 15 | 17
Completed (Total number of participants (adolescents and caregivers) completed) | 25 | 26
Not Completed | 0 | 1
Not completed — Excluded from analyses | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (Control) | FP Decision Tool and Discussion (Treatment) | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Full Range); unit: Mean] — Age Population: Rows refer to the number of specific participant types (adolescents and caregivers separately) whereas the Overall number refers to the number of participants combined. As a note, discrepancies between baseline characteristics and participant flow are attributed to missing data/skipped questions.
  Mean
    Adolescents: number analyzed (Participants) | 10 | 9 | 19
    Adolescents | 17 [14 to 24] | 17 [14 to 24] | 17 [14 to 24]
    Caregivers: number analyzed (Participants) | 15 | 13 | 28
    Caregivers | 46 [36 to 65] | 44 [36 to 55] | 45 [36 to 65]
    Overall: number analyzed (Participants) | 25 | 22 | 47
    Overall | 33 [14 to 65] | 31 [14 to 55] | 32 [14 to 65]
Sex: Female, Male [Count of Participants; unit: Participants] — Biological Sex (for adolescents, only biological males were deemed eligible) Population: Rows refer to the number of specific participant types (adolescents and caregivers separately) whereas the Overall number refers to the number of participants combined. As a note, discrepancies between baseline characteristics and participant flow are attributed to missing data/skipped questions.
  Participants
    Adolescents: number analyzed (Participants) | 10 | 9 | 19
    Adolescents: Female | 0 | 0 | 0
    Adolescents: Male | 10 | 9 | 19
    Caregivers: number analyzed (Participants) | 15 | 17 | 32
    Caregivers: Female | 12 | 9 | 21
    Caregivers: Male | 3 | 8 | 11
    Overall: Female | 12 | 9 | 21
    Overall: Male | 13 | 17 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity Population: Rows refer to the number of specific participant types (adolescents and caregivers separately) whereas the Overall number refers to the number of participants combined.
  Participants
    Adolescents: number analyzed (Participants) | 10 | 9 | 19
    Adolescents: Hispanic or Latino | 0 | 0 | 0
    Adolescents: Not Hispanic or Latino | 9 | 9 | 18
    Adolescents: Unknown or Not Reported | 1 | 0 | 1
    Caregiver: number analyzed (Participants) | 15 | 17 | 32
    Caregiver: Hispanic or Latino | 1 | 1 | 2
    Caregiver: Not Hispanic or Latino | 14 | 16 | 30
    Caregiver: Unknown or Not Reported | 0 | 0 | 0
    Overall: Hispanic or Latino | 1 | 1 | 2
    Overall: Not Hispanic or Latino | 23 | 25 | 48
    Overall: Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race Population: Rows refer to the number of specific participant types (adolescents and caregivers separately) whereas the Overall number refers to the number of participants combined.
  Participants
    Adolescents: number analyzed (Participants) | 10 | 9 | 19
    Adolescents: American Indian or Alaska Native | 0 | 0 | 0
    Adolescents: Asian | 0 | 1 | 1
    Adolescents: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Adolescents: Black or African American | 0 | 0 | 0
    Adolescents: White | 9 | 8 | 17
    Adolescents: More than one race | 0 | 0 | 0
    Adolescents: Unknown or Not Reported | 1 | 0 | 1
    Caregivers: number analyzed (Participants) | 15 | 17 | 32
    Caregivers: American Indian or Alaska Native | 1 | 0 | 1
    Caregivers: Asian | 0 | 2 | 2
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers: Black or African American | 1 | 1 | 2
    Caregivers: White | 12 | 11 | 23
    Caregivers: More than one race | 1 | 3 | 4
    Caregivers: Unknown or Not Reported | 0 | 0 | 0
    Overall: American Indian or Alaska Native | 1 | 0 | 1
    Overall: Asian | 0 | 3 | 3
    Overall: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Overall: Black or African American | 1 | 1 | 2
    Overall: White | 21 | 19 | 40
    Overall: More than one race | 1 | 3 | 4
    Overall: Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Fertility Preservation (FP) Uptake
Description: Fertility Preservation (FP) Uptake (measured by the number of adolescents/adolescents of caregivers who attempted FP)
Time Frame: Baseline to before AYA begins treatment (generally within one to two weeks from baseline)
Population: As a note, discrepancies between baseline characteristics and participant flow are attributed to missing data/skipped questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (Control) | FP Decision Tool and Discussion (Treatment)
Number analyzed (Participants) | 10 | 9
Participants | 10 | 9
Statistical Analysis 1: Comparison: Standard of Care (Control) vs FP Decision Tool and Discussion (Treatment); Chi-square test was used to determine if study arm is associated with FP uptake; Test type: Other — Chi-squared test was used to determine if study arm is associated with FP uptake; p = .64, Chi-squared; df=(1, 19)

2. Secondary Outcome: Brief Subjective Decision Quality (BSDQ) Questionnaire - AYA
Description: AYAs will complete the six-item Brief Subjective Decision Quality (BSDQ) Questionnaire with total scores ranging from 1-7; higher scores indicate more satisfaction with their decision.
Time Frame: 1-month post randomization
Population: These analyses were conducted on each BSDQ item by participant type (adolescents and caregivers). Some participants skipped questions resulting in differences in "n" values by each item. Some participants did not complete this 1-month post randomization visit.
Measure: Mean (Standard Deviation); unit: Mean
Arm/Group | Standard of Care (Control) | FP Decision Tool and Discussion (Treatment)
Number analyzed (Participants) | 9 | 9
Mean
  Adolescent BSDQ Regret Mean: number analyzed (Participants) | 8 | 9
  Adolescent BSDQ Regret Mean | 1.9 (1.6) | 1.0 (0.0)
  Adolescent BSDQ Satsifaction Mean: number analyzed (Participants) | 8 | 9
  Adolescent BSDQ Satsifaction Mean | 5.9 (1.4) | 5.3 (2.5)
  Adolescent BSDQ Information Mean: number analyzed (Participants) | 8 | 9
  Adolescent BSDQ Information Mean | 6.3 (1.0) | 6.3 (1.0)
  Adolescent BSDQ Time Mean | 4.6 (2.6) | 6.3 (1.0)
  Adolescent BSDQ Involvement Mean | 6.1 (1.5) | 6.8 (0.7)
  Adolescent BSDQ "Right for You" Mean | 3.9 (2.5) | 5.4 (1.4)

3. Secondary Outcome: Brief Subjective Decision Quality (BSDQ) Questionnaire - Caregiver
Description: Caregivers will complete the six-item Brief Subjective Decision Quality (BSDQ) Questionnaire with total scores ranging from 1-7; higher scores indicate more satisfaction with their decision.
Time Frame: 1-month post randomization
Population: Some participants skipped individual items. Some participants did not complete this 1-month post randomization visit.
Measure: Mean (Standard Deviation); unit: Mean
Arm/Group | Standard of Care (Control) | FP Decision Tool and Discussion (Treatment)
Number analyzed (Participants) | 11 | 14
Mean
  Caregiver BSDQ Regret: number analyzed (Participants) | 11 | 13
  Caregiver BSDQ Regret | 2.6 (2.2) | 1.4 (1.0)
  Caregiver BSDQ Satisfaction: number analyzed (Participants) | 11 | 13
  Caregiver BSDQ Satisfaction | 5.6 (2.0) | 5.7 (2.2)
  Caregiver BSDQ Information | 5.7 (2.1) | 5.7 (2.0)
  Caregiver BSDQ Time | 4.5 (2.4) | 5.1 (1.5)
  Caregiver BSDQ Involvement | 5.5 (2.4) | 5.7 (2.0)
  Caregiver BSDQ "Right for you": number analyzed (Participants) | 11 | 11
  Caregiver BSDQ "Right for you" | 5.5 (2.1) | 5.0 (1.9)

4. Secondary Outcome: Brief Subjective Decision Quality (BSDQ) Questionnaire - AYA
Description: as for outcome 2
Time Frame: 1-year post randomization
Population: These analyses were conducted on each BSDQ item by participant type (adolescents and caregivers). Some participants skipped questions resulting in differences in "n" values by each item. Some participants did not complete this 1-year post randomization visit.
Measure: Mean (Standard Deviation); unit: Mean
Arm/Group | Standard of Care (Control) | FP Decision Tool and Discussion (Treatment)
Number analyzed (Participants) | 9 | 9
Mean
  Adolescent BSDQ Regret | 1.7 (1.0) | 1.1 (0.3)
  Adolescent BDSQ Satisfaction | 5.7 (1.4) | 6.0 (1.5)
  Adolescent BSDQ Information | 6.1 (2.0) | 6.3 (2.0)
  Adolescent BSDQ Time | 5.7 (2.0) | 6.3 (1.4)
  Adolescent BSDQ Involvement | 6.5 (1.4) | 5.9 (2.0)
  Adolescent BSDQ "Right for you" | 4.6 (1.7) | 5.7 (1.7)

5. Secondary Outcome: Brief Subjective Decision Quality (BSDQ) Questionnaire - Caregiver
Description: as for outcome 3
Time Frame: 1-year post randomization
Population: Some participants skipped individual items. Some participants did not complete this 1-year post randomization visit.
Measure: Mean (Standard Deviation); unit: Mean
Arm/Group | Standard of Care (Control) | FP Decision Tool and Discussion (Treatment)
Number analyzed (Participants) | 8 | 9
Mean
  Caregiver BSDQ Regret | 1.8 (1.4) | 1.4 (1.0)
  Caregiver BSDQ Satisfaction | 5.4 (1.8) | 5.9 (2.1)
  Caregiver BSDQ Information | 6.5 (0.9) | 7.0 (0.0)
  Caregiver BSDQ Time | 3.8 (2.6) | 4.8 (1.9)
  Caregiver BSDQ Involvement | 6.8 (0.7) | 5.9 (1.8)
  Caregiver BSDQ "Right for you" | 4.3 (1.6) | 5.1 (2.1)

ADVERSE EVENTS:
Time Frame: Approximately four years (from enrollment to present since data collection is ongoing)
Description: Caregiver and adolescent dyads were randomized as a group, but adverse events were reported separately for each participant type.
Groups:
- Standard of Care (Control) - Adolescent; Standard of Care (Control) - Caregiver: Participants will receive a standard of care fertility consult.
- FP Decision Tool and Discussion (Treatment) - Adolescent; FP Decision Tool and Discussion (Treatment) -Caregivers: Participants will receive a standard of care fertility consult and will participate in a family-centered psychoeducational intervention consisting of completing a FP Decision Tool and participating in a guided discussion about responses and discrepancies identified in the FP Decision Tool.
  FP Decision Tool and Discussion: The intervention will be administered by a trained interventionist. The interventionist will administer the digital FP Decision Tool to families in the intervention arm. The tool asks questions examining each AYA's thoughts or feelings regarding parenthood and fertility preservation. The parent version asks the same questions, plus additional questions asking the parent to rate their son's feelings on certain topics (i.e., whether their son wants to have a child, whether their son would be as happy with an adopted child versus a biological child). Items are coded based on the domains of the Health Belief Model (perceived benefits, perceived barriers, perceived threats, self-efficacy, and cues to action). Items are scored and the trained interventionist will facilitate a guided discussion based on the family's responses and discrepancies.
Arm/Group | Standard of Care (Control) - Adolescent | FP Decision Tool and Discussion (Treatment) - Adolescent | Standard of Care (Control) - Caregiver | FP Decision Tool and Discussion (Treatment) -Caregivers
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT04268004/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT04268004/ICF_001.pdf